CLINICAL TRIAL: NCT06737055
Title: The Dream Team: Testing Implementation of a Sleep Intervention for Perinatal Women Delivered by Direct Care Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Bradley Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1848819
Record Dates: First submitted 2024-07-01; First posted 2024-12-17 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Sleep; Postpartum Depression; Pregnancy Related; Insomnia; Sleep Deprivation; Sleep Hygiene; Sleep Disturbance
Keywords: Home visitors; sleep diaries; education; implementation; RE-AIM
MeSH Terms: conditions — Depression, Postpartum; Sleep Initiation and Maintenance Disorders; Sleep Deprivation; Sleep Hygiene; Parasomnias

STUDY DESIGN:
Intervention Model Description: This is an implementation science project to develop and test an educational program for teaching home visitors and expectant and new parents about sleep. The study uses the RE-AIM framework.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Visitors (Experimental): The participants in Phase 1 of the proposed study are individuals who provide services to perinatal women who are at risk of postpartum depression. The investigators will recruit 35 adults ages 18 years or older who provide health, well-being, and/or mental health services/treatment to pregnant and postpartum women to participate in Phase 1 of this study. Job titles that meet inclusion criteria include nurses, nurse practitioners, family support workers, therapists, counselors, doulas, lactation consultants, childbirth educators, social workers, public health workers, midwives, and nurse midwives. The investigators will not select participants based on age, gender, sex, or racial or ethnic identity.
  Interventions: Behavioral: Education about behavioral strategies to improve sleep
- Expectant and New Parents (Experimental): Phase 2 participants will be given access to the educational materials about sleep and the investigators will collect information about their sleep.
  To qualify for enrollment, Phase 2 participants must be:
  * expectant parents OR new parents up to 1 year postpartum
  * 18 to 45 years old
  * receiving community-based health, well-being, and or mental health services or treatment from individuals who participated in Phase 1
  * speak and read English or Spanish
  * have access to a smart phone to view the training videos and complete the sleep diaries and assessments
  * are experiencing clinically significant sleep difficulties defined as an Insomnia Severity Index score greater than 7 The investigators will exclude potential participants who are parents whose infants will not be living in the home or who will have a nighttime caregiver
  Interventions: Behavioral: Education about behavioral strategies to improve sleep

INTERVENTIONS:
Behavioral: Education about behavioral strategies to improve sleep — In collaboration with direct care workers, the investigators are developing an intervention to help home visitors support clients who experience sleep difficulties in the perinatal period. The intervention consists of a series of educational videos about promoting healthy sleep and addressing sleep difficulties during pregnancy and the postpartum period.
  Other Names: Dream Team Training

SUMMARY:
Insufficient and disrupted sleep are rarely addressed in expectant and new mothers, despite evidence that disturbed sleep is a modifiable risk factor for negative health outcomes for mothers and their children. In this study the investigators will adapt, refine, and pilot test the implementation of a behavioral sleep intervention consisting of short videos designed to accompany a free behavioral sleep app. In Phase 1, the investigators will develop and refine the intervention with input from direct care workers who serve at-risk perinatal women. In Phase 2, direct care workers will deploy the training to expectant mothers with sleep concerns and the investigators will assess the reach, effectiveness, adoption, implementation, and maintenance of this scalable, efficient intervention to improve sleep.

DETAILED DESCRIPTION:
Disrupted, insufficient sleep occurs in the majority of pregnant women and increases the risk of negative health consequences for mothers and their infants, including pregnancy and childbirth complications as well as chronic illnesses, such as major depression and weight retention/obesity. Conventionally, perinatal sleep disturbances have been viewed as expected and intractable, but recent studies demonstrate that behavioral interventions are effective for improving sleep in pregnant and postpartum women. Nevertheless, efficient, scalable sleep interventions that are tailored to expectant and new mothers are scarce. This Administrative Supplement for Research on Women's Health seeks to develop a high-fidelity, evidence-based sleep intervention in collaboration with direct care workers who engage with perinatal women and to collect preliminary data regarding delivery of the resulting intervention to expectant and new parents. This pilot project is grounded in the RE-AIM framework, and will assess the Reach, Effectiveness, Adoption, Implementation, and Maintenance dimensions of this model to prepare for a large-scale future R01 hybrid effectiveness-implementation trial. In Phase 1, the investigators will develop short, evidence-based, educational videos in English (with Spanish subtitles) that focus on improving perinatal sleep and that map onto modules in the free, publicly-available mobile app, CBTi Coach. Videos will be produced and refined in cooperation with direct care workers and a video production company with community engagement experience. Direct care workers who work with perinatal women will be trained to deliver the intervention (target n=35). In Phase 2, direct care workers will be invited to use the intervention with clients who report sleep problems and the investigators will study implementation in workers and clients (target n=20).

ELIGIBILITY:
Phase 1 Inclusion Criteria:

To qualify for Phase 1 enrollment, participants must be:

* over 18 years of age;
* working with expectant and new mothers in a community setting (i.e., outpatient clinic, social service agency, home visiting program, community center);
* in a role where they would be expected to meet with the same client on at least 4 occasions during the perinatal period; in situations where a team-based approach is used to provide services and a client may not see the exact same person at each visit, team members will qualify if they all enroll in the study (e.g., two nurse midwives who provide coverage for each other may both enroll);
* have access to a smart phone to view the training videos, complete the assessments, and access the free CBTi Coach app; speak and read English or Spanish;
* express interest in providing their clients with additional tools to manage sleep disturbances in pregnancy and the postpartum period.

Phase 1 Exclusion Criteria:

The investigators will exclude potential participants who:

* already have certification or a specialty in perinatal sleep (e.g., therapists with formal training in CBTi, individuals with sleep coaching practices);
* those who do not have longitudinal relationships with clients (e.g., intake workers).

Phase 2 Inclusion Criteria:

To qualify, Phase 2 participants must be:

* expectant parents OR new parents up to 1 year postpartum;
* age 18 to 45 years old;
* receiving community-based health, well-being, and or mental health services or treatment from individuals who participated in Phase 1;
* speak and read English or Spanish;
* have access to a smart phone to view the training videos and complete the assessments;
* have clinically significant sleep difficulties defined as an Insomnia Severity Index score greater than 7.

Phase 2 Exclusion Criteria:

The investigators will exclude potential participants whose infants will not be living in the home or who will have a nighttime caregiver.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Reach | Throughout training period, i.e., for about 6 months; one time measure.
  Reach: Number of eligible workers who enroll in the training and number of workers who complete the training
Phase 1 Effectiveness | At enrollment and 1 month after training.
  Effectiveness: Participants are tested before and after training on sleep and circadian rhythm knowledge. Questions are based on the learning objectives for the educational modules. A successful outcome will be defined as >= 70% of sleep knowledge questions answered correctly.
Phase 1 Acceptability | 1 month after training
  Acceptability: Participants will complete an online questionnaire to assess their perceptions of the training videos including Likert scales where they will report on (a) how prepared they feel to deliver the intervention; (b) ease of use; (c) compatibility with other resources they provide; and (d) the likelihood that they will use the app with their clients. This questionnaire will also include a short answer section for participants to report facilitators and barriers to use of the intervention.
Phase 2 Reach | one time measure during enrollment period, ~ 6 months
  Reach: Investigators will track what percent of clients who are referred actually enroll, the number of pregnant vs. postpartum women who enroll, and the number of fathers/partners who enroll.
Phase 2 Effectiveness | 6 weeks after enrollment
  Effectiveness: Clients will complete a brief survey to assess their perceptions of the acceptability and utility of the intervention.
Phase 2 Effectiveness - Insomnia Severity Index | at enrollment and 6 weeks after enrollment
  Participants will complete the 7-item Insomnia Severity Index (ISI, range 0-28, higher scores indicate more sleep disturbance) at enrollment and 6 weeks after enrollment.
Phase 2 Effectiveness - Implementation | from enrolllment through 6 weeks after enrollment
  Implementation: After clients enroll, investigators will assess quantitative implementation measures related to whether clients engage with the intervention as intended through metadata provided by the app and website (i.e., time spent on the app in minutes and time spent viewing videos in minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Sharkey, MD, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
The final computerized research datasets will include both raw and summary data as well as documentation so that others can make use of the data. These data represent a valuable public resource and the investigators strongly support the notion that other researchers will be able to capitalize on the efforts and funding that go into collecting and processing these data.
Supporting Information: Study Protocol, ICF
Time Frame: The informed consent documents will be posted on a federal website after enrollment closes and no later than 60 days after the last study visit of any participant. English language consent forms will be posted at ClinicalTrials.gov and Non-English consent forms will be posted to Regulations.gov. Additionally, results will be reported no later than one year after the actual completion date listed in ClinicalTrials.gov.
Access Criteria: By request to the PI.

DOCUMENTS (1):
  • Informed Consent Form (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT06737055/ICF_000.pdf